CLINICAL TRIAL: NCT03442114
Title: Engaging Parents of Children With Sickle Cell Anemia and Their Providers in Shared-Decision Making for Hydroxyurea (ENGAGE HU)
Brief Title: Shared-Decision Making for Hydroxyurea
Acronym: ENGAGE-HU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CDR_1609_36055
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Anemia; Children, Only
Keywords: shared decision making; parent-provider communication; hydroxyurea; sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxyurea SDM Toolkit (H-SDM) (Experimental): During the H-SDM toolkit condition, sites will develop methods for identifying Eligible Patients & Monitoring Progress, have the opportunity to use Implementation Tools, and will use the Visit Decision Aids. The H-SDM toolkit has four visit decision aids to support parents in their decision about hydroxyurea: pre-visit brochure, in-visit issue card, after-visit booklet and video narratives {videos of parents telling their story about how they made a decision about hydroxyurea).
  Interventions: Behavioral: Hydroxyurea SDM Toolkit
- Clinician Pocket Guide (Active Comparator): In this condition, sites will provide current guidelines for offering hydroxyurea and use the American Society of Hematology (ASH) pocket guide as a reference. ASH developed 'The Hydroxyurea and Transfusion Therapy for the Treatment of Sickle Cell Disease' clinician pocket guide based on the National Heart, Lung, and Blood Institute's Evidence Based Management of Sickle Cell Disease: Expert Panel Report, 2014.'
  Interventions: Behavioral: Clinician Pocket Guide

INTERVENTIONS:
Behavioral: Hydroxyurea SDM Toolkit — Implementation tools and visit decision aids
  Arms: Hydroxyurea SDM Toolkit (H-SDM)
Behavioral: Clinician Pocket Guide — current hydroxyurea protocol and ASH pocket guide
  Arms: Clinician Pocket Guide

SUMMARY:
The goal of the study is to understand how best to help parents of young children with sickle cell disease and their clinicians have a shared discussion about hydroxyurea (one that takes into account medical evidence and parent values and preferences). The study will compare two methods to help clinicians facilitate this-a clinician pocket guide and a clinician hydroxyurea shared decision making toolkit-in a group of parents of children ages 0-5 with sickle cell disease. The investigators hope that both methods lead to parents reaching a high-quality, well-informed decision. In addition, the team hopes to demonstrate that parents who experience a shared decision will have lower anxiety and decisional uncertainty. The researchers also expect these parents to be more likely to choose hydroxyurea and that their children will have less pain, fewer hospitalizations, better developmental outcomes, and higher quality of life. The project team hopes to show that the toolkit method is easy for clinicians to use and gives parents the support needed to make an informed decision.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a genetic blood disorder that places children at risk for serious medical complications, early morbidity and mortality, and high healthcare utilization. In the U.S., SCD primarily affects African-American and Latino children. Hydroxyurea is one of the only disease-modifying treatment for this devastating and life-threatening disease. National Evidence-Based Guidelines recommend the use of a shared decision making approach to offer hydroxyurea to all children with SCD as early as nine months of age. Hydroxyurea uptake remains low because parents lack information about hydroxyurea and have concerns about its safety and potential long-term side effects (e.g. cancer, infertility, birth defects). Clinicians do not have the training or tools to facilitate a shared discussion with parents that provides medical evidence and considers parent preferences and values. The current study compares two methods for disseminating hydroxyurea guidelines and facilitating shared decision-making: the American Society of Hematology's hydroxyurea clinician pocket guide (usual care method) and a clinician hydroxyurea shared decision-making toolkit (H-SDM toolkit). The specific aims of the study are to evaluate the effectiveness of the usual care dissemination method (clinician pocket guide) and the H-SDM clinician toolkit dissemination method on: parent report of decisional uncertainty (primary outcome chosen by parents of children with SCD), parent perception of experiencing shared decision-making, parent knowledge of hydroxyurea, the number of children offered hydroxyurea, hydroxyurea uptake (those with active prescriptions), and child health outcomes (pain, neurocognitive functioning, sickle cell related quality of life and healthcare utilization). Eligible children must be between the ages of 0 and 5 and a candidate for hydroxyurea to participate. The trial will use a stepped-wedge design (clinic is the unit of randomization). The long-term objective of the research team is to improve the quality of care for children with SCD. The investigators propose that suboptimal care for patients with SCD is preventable with the use of multicomponent dissemination methods if developed with key stakeholders and designed to address barriers to high quality care at multiple levels (patient, clinician, healthcare system, and community).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: sickle cell disease
2. Age: birth-5 years, inclusive
3. Eligible for hydroxyurea (genotype SS, Sβ0Thal or other genotype + clinical complications)
4. Child's parent, legal guardian, or designated decision maker (caregiver) must participate in both study visits
5. Child's parent, legal guardian, or designated decision maker (caregiver) must able to read, understand, and speak English

Exclusion Criteria:

1. Parent/legal guardian has previously been approached OR made a decision about whether to initiate hydroxyurea.
2. Any and all other diagnoses or conditions which, in the opinion of the site investigator or hematologist, would prevent the patient from being a suitable candidate for the study.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori E Crosby, PsyD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (11):
- United States (11):
  - UCSF Beinoff Children's Hospital and Research Center at Oakland, Oakland, California
  - Nemours Children's Health, Wilmington, Delaware
  - Howard University, Washington D.C., District of Columbia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - The Washington University, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
This study will comply with the Patient Centered Outcomes Research Institute (PCORI) Public Access Policy, which ensures that the public has access to the published results of PCORI funded research.

REFERENCES:
- [Derived] Williford DN, McTate EA, Hood AM, Reader SK, Hildenbrand AK, Smith-Whitley K, Creary SE, Thompson AA, Hackworth R, Raphael JL, Crosby LE. Psychologists as leaders in equitable science: Applications of antiracism and community participatory strategies in a pediatric behavioral medicine clinical trial. Am Psychol. 2023 Feb-Mar;78(2):107-118. doi: 10.1037/amp0001086. PMID 37011163
- [Derived] Strong H, Hood AM, Johnson Y, Hackworth R, Reed-Shackelford M, Ramaswamy R, Varughese T, Quinn CT, Crosby LE. Using the consolidated framework for implementation research to identify recruitment barriers and targeted strategies for a shared decision-making randomized clinical trial in pediatric sickle cell disease. Clin Trials. 2023 Jun;20(3):211-222. doi: 10.1177/17407745231154199. Epub 2023 Feb 16. PMID 36794731
- [Derived] Hood AM, Strong H, Nwankwo C, Johnson Y, Peugh J, Mara CA, Shook LM, Brinkman WB, Real FJ, Klein MD, Hackworth R, Badawy SM, Thompson AA, Raphael JL, Yates AM, Smith-Whitley K, King AA, Calhoun C, Creary SE, Piccone CM, Hildenbrand AK, Reader SK, Neumayr L, Meier ER, Sobota AE, Rana S, Britto M, Saving KL, Treadwell M, Quinn CT, Ware RE, Crosby LE. Engaging Caregivers and Providers of Children With Sickle Cell Anemia in Shared Decision Making for Hydroxyurea: Protocol for a Multicenter Randomized Controlled Trial. JMIR Res Protoc. 2021 May 21;10(5):e27650. doi: 10.2196/27650. PMID 34018965

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Since children were 0-5 years of age, parents completed all measures and were considered study participants. Study participants were recruited based on how they met inclusion criteria assessed by Clinical Research Coordinators and approved by participating physicians at 12 academic medical centers between July 2018 and November 2021.
Pre-assignment Details: This study was originally designed as a stepped-wedge cluster randomized trial design. However, the study was amended to randomize participants instead of facilities, resulting in a parallel randomized controlled clinical trial.
  Of 176 enrolled participants,174 were allocated to either the Usual Care or Toolkit condition (quasi-experimental design), but only 137 completed the study. While parents completed the surveys and provided feedback, only children were enrolled in the study.
Groups:
- Hydroxyurea Shared Decision Making Toolkit (H-SDM): During the H-SDM toolkit condition, sites will develop methods for identifying Eligible Patients & Monitoring Progress, have the opportunity to use Implementation Tools, and will use the Visit Decision Aids. The H-SDM toolkit has four visit decision aids to support parents in their decision about hydroxyurea: pre-visit brochure, in-visit issue card, after-visit booklet and video narratives {videos of parents telling their story about how they made a decision about hydroxyurea).
  Hydroxyurea SDM Toolkit: Implementation tools and visit decision aids
Period: Overall Study
Arm/Group | Hydroxyurea Shared Decision Making Toolkit (H-SDM) | Clinician Pocket Guide
Started | 94 | 80
Completed | 78 | 59
Not Completed | 16 | 21
Not completed — Lost to Follow-up | 13 | 13
Not completed — Physician Decision | 2 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Guardianship Change | 0 | 1

BASELINE CHARACTERISTICS:
Population: These numbers represent 292 unique participants. 83 children and 83 parents in the Clinician Pocket Guide Arm and 63 children and 63 parents in the Hydroxyurea SDM Toolkit (H-SDM) Arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinician Pocket Guide | Hydroxyurea SDM Toolkit (H-SDM) | Total
Number analyzed (Participants) | 166 | 126 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] — Age as calculated using date of birth and date of visit. Population: Baseline measure stratified into parents and children.
  years
    Parent/Guardian: number analyzed (Participants) | 83 | 63 | 146
    Parent/Guardian | 30.00 (6.891) | 30.32 (7.980) | 30.13 (7.345)
    Child: number analyzed (Participants) | 83 | 63 | 146
    Child | 1.05 (1.333) | 1.20 (1.547) | 1.11 (1.425)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data not collected for one child and one parent in the "H-SDM" Arm.
  Participants
    Parent/Guardian: number analyzed (Participants) | 83 | 62 | 145
    Parent/Guardian: Female | 76 | 60 | 136
    Parent/Guardian: Male | 7 | 2 | 9
    Child: number analyzed (Participants) | 83 | 62 | 145
    Child: Female | 45 | 32 | 77
    Child: Male | 38 | 30 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline measure stratified into parents and children.
  Participants
    Parent/Guardian: number analyzed (Participants) | 83 | 63 | 146
    Parent/Guardian: American Indian or Alaska Native | 0 | 0 | 0
    Parent/Guardian: Asian | 0 | 1 | 1
    Parent/Guardian: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent/Guardian: Black or African American | 74 | 56 | 130
    Parent/Guardian: White | 1 | 1 | 2
    Parent/Guardian: More than one race | 6 | 3 | 9
    Parent/Guardian: Unknown or Not Reported | 2 | 2 | 4
    Child: number analyzed (Participants) | 83 | 63 | 146
    Child: American Indian or Alaska Native | 0 | 0 | 0
    Child: Asian | 0 | 0 | 0
    Child: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Child: Black or African American | 79 | 57 | 136
    Child: White | 0 | 1 | 1
    Child: More than one race | 4 | 4 | 8
    Child: Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 166 | 126 | 292

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict
Description: Decisional Conflict Scale (DCS) is a 16-item parent-completed survey that measures uncertainty experienced when feeling uninformed about options, unclear about personal values, or unsupported in making a choice. Parents report their level of agreement with each item using a 5 point likert scale (0=strongly agree to 4=strongly disagree). For the total score, items are summed, divided by 16, and multiplied by 25. All subscores consist of 3 items except the Effective Decisions subcore (4 items) that are summed, divided by the number of items (3 or4) and multiplied by 25.
  Scores range from 0 (feels extremely certain about best choice) to 100 (feels extremely uncertain about best choice) on the total score and all subscores. Thus, a higher score indicates a high decisional conflict.
Time Frame: Baseline - after shared discussion with clinician
Population: All parents with data for baseline measures (146) were included in the analyses, whether or not they attended the follow-up visit or completed additional measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Pocket Guide | Hydroxyurea SDM Toolkit (H-SDM)
Number analyzed (Participants) | 83 | 63
score on a scale
  DCS Total Score | 22.9 (20.3) | 19.8 (17.1)
  Uncertainty | 26.9 (25.4) | 23.5 (21.5)
  Informed | 20.8 (20.2) | 16.8 (14.4)
  Values Clarity | 23.3 (24.4) | 21.0 (21.1)
  Support | 21.2 (24.4) | 17.9 (16.8)
  Effective Decisions | 22.3 (21.0) | 19.6 (20.3)

2. Primary Outcome: Dyadic OPTION
Description: Dyadic OPTION describes clinician behaviors to involve a patient/parent in decision-making. A total score is calculated which ranges from 0 (no involvement) to 100 (maximal involvement). Dyadic OPTION scores correlate well with OPTION scale (Melbourne et al., 2011); 1 item "My doctor and I made the decision together"(Légaré et al., 2010). Higher scores indicate that the patient/parent has higher shared decision making competencies.
Time Frame: Baseline visit - after shared discussion with clinician
Population: 145 parents with data for baseline measures were included in the analyses whether or not they attended the follow-up visit or completed additional measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Pocket Guide | Hydroxyurea SDM Toolkit (H-SDM)
Number analyzed (Participants) | 82 | 63
score on a scale | 39.8 (6.7) | 40.3 (5.8)

3. Secondary Outcome: Hydroxyurea Offered
Description: 1 of 3 responses - completed by the research coordinator based on review of electronic medical record (EMR) data: hydroxyurea was not offered, offered, or previously prescribed.
Time Frame: From date of randomization until the date of first documented offering or prescription, whichever came first, assessed up to 7 months
Population: 143 children with data for baseline measures were included in the analyses whether or not they attended the follow-up visit or completed additional measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Pocket Guide | Hydroxyurea SDM Toolkit (H-SDM)
Number analyzed (Participants) | 83 | 60
Participants
  Offered | 61 | 32
  Not Offered | 19 | 25
  Previously Prescribed | 3 | 3

4. Secondary Outcome: Satisfaction With Decision-Making
Description: Eight-item survey adapted from the Satisfaction With Decision scale 41 (4 items) and the Agency for Healthcare Research and Quality's Consumer Assessment of Healthcare Providers and Systems survey related to patient experience of care (4 items). 42 Items are summed to obtain a total score ranging from 0 to 28, with higher scores indicating higher satisfaction.
Time Frame: Baseline after the shared discussion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Pocket Guide | Hydroxyurea SDM Toolkit (H-SDM)
Number analyzed (Participants) | 82 | 63
score on a scale | 13.5 (5.5) | 13.2 (6.3)

5. Secondary Outcome: Ages & Stages Questionnaire - Gross Motor Subscale
Description: This questionnaire is a reliable, accurate developmental and social-emotional screener for children between birth and 6 years of age, with a Cronbach α = .60 to .85. Scores range from 0 to 60, with higher scores indicating that the child's development is on schedule.
Time Frame: After discussion with clinician
Population: The data of 120 children with baseline measures were included in the analyses whether or not they attended the follow-up visit or completed additional measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Pocket Guide | Hydroxyurea SDM Toolkit (H-SDM)
Number analyzed (Participants) | 75 | 45
score on a scale | 50.9 (14.0) | 51.9 (11.0)

6. Secondary Outcome: Pediatric Quality of Life Inventory - Sickle Cell Disease Module (Peds QL - SCD Module) - Total Score
Description: Parent report of sickle cell disease (SCD)-specific quality of life (QOL) and pain, as measured by the Pediatric Quality of Life (PedsQL) SCD Module, which assesses several domains of health-related quality of life (HRQOL), including pain impact, fatigue, pain management, emotions, communication, and treatment adherence. Scores range from 0 to 100, with higher scores indicating higher HRQOL or higher functioning.
Time Frame: After shared discussion with clinician
Population: 121 children with data for baseline measures were included in the analyses whether or not they attended the follow-up visit or completed additional measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Pocket Guide | Hydroxyurea SDM Toolkit (H-SDM)
Number analyzed (Participants) | 74 | 47
score on a scale | 82.5 (15.5) | 82.0 (15.5)

7. Secondary Outcome: Hydroxyurea Knowledge
Description: Eight-item survey developed based on the existing literature, the Ottawa Knowledge User Manual, and parent and clinician stakeholders and used in our pilot work. Items are summed to obtain a total score ranging from 0 to 9, with higher scores indicating more knowledge.
Time Frame: After shared discussion with clinician
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Pocket Guide | Hydroxyurea SDM Toolkit (H-SDM)
Number analyzed (Participants) | 82 | 63
score on a scale | 6.3 (1.7) | 6.1 (1.5)

ADVERSE EVENTS:
Time Frame: Clinical Research Coordinators reported any adverse event data that occurred for the child with sickle cell disease enrolled between baseline and follow-up visits, which took place anywhere between 3 to 7 months. Numbers reported are based on all children enrolled in the overall study, not just those with data available for analyses (n=146).
Description: An adverse events survey was filled out by each participating site's Clinical Research Coordinator(s) during the follow-up visit. Mortality and Adverse Events were not monitored/assessed in the parent population.
Arm/Group | Clinician Pocket Guide | Hydroxyurea SDM Toolkit (H-SDM)
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/80
Serious Adverse Events (participants affected / at risk) | 5/94 | 1/80
Other Adverse Events (participants affected / at risk) | 3/94 | 2/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinician Pocket Guide (N=94) | Hydroxyurea SDM Toolkit (H-SDM) (N=80)
Hospitalization (Blood and lymphatic system disorders) | 5 (5) | 1 (1) — Hospitalization due to patient condition/disorder; not related to intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinician Pocket Guide (N=94) | Hydroxyurea SDM Toolkit (H-SDM) (N=80)
Emergency Department (ED) Visit (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Emergency Department/Room Visit due to participant condition/disorder; not related to intervention
ED visit for Vasoocclusive Sickle Cell Crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — ED visit for Vasoocclusive Sickle Cell Crisis related to patient condition/disorder; not related to intervention
Hospitalization (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Hospitalization due to patient condition/disorder; not related to intervention

LIMITATIONS AND CAVEATS:
Due to challenges with study implementation, low accrual, and COVID-19, the study design was changed from a stepped wedge to a quasi-experimental observational study. We were able to maintain some of the advantages of the stepped wedge including that all sites received the Toolkit dissemination method. We also considered site and cluster effects in our analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03442114/Prot_SAP_002.pdf
  • Informed Consent Form (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT03442114/ICF_001.pdf